CLINICAL TRIAL: NCT00458263
Title: One Arm, Open Study to Assess Biochemical Markers of Growth Response to Growth Hormone Treatment in Children With Idiopathic Short Stature
Brief Title: Biochemical Markers of Growth Response to Growth Hormone Treatment in Children With Idiopathic Short Stature
Acronym: ISS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: rmc003515ctil
Record Dates: First submitted 2007-04-08; First posted 2007-04-10 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2011-10

CONDITIONS: Idiopathic Short Stature
Keywords: Growth Hormone treatment; ISS; Biochemical markers; Growth response

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- single arm (Experimental)
  Interventions: Drug: Somatotropin growth hormone recombinant human

INTERVENTIONS:
Drug: Somatotropin growth hormone recombinant human — daily Sub Cutaneous injections

SUMMARY:
One arm, open, prospective, intervention study to assess biochemical markers of growth response to Growth Hormone treatment in 20 Children, aged 3-9 years old, with idiopathic short stature. All participants will be treated with Growth Hormone during the first year of the study (and then in accordance with the local ethic requirement, to supply drug which is not approved for the indication used in the study, for additional 3 years) and then will be followed up for the next 3 years. The impact of Growth Hormone therapy on clinical laboratory parameters that are indicative of the growth response will be assessed by collecting blood and urine samples during the 4 years study period. The primary endpoints are measurements of height and growth velocity during the year of Growth Hormone treatment, the height at the beginning of puberty and final height. Secondary endpoints are psychological parameters, assessed by questionnaires.

DETAILED DESCRIPTION:
One arm, open prospective intervention study to assess biochemical markers of growth response to Growth Hormone treatment in 20 children, aged 3-9 years old, with idiopathic short stature.

Objectives:

1. To determine axiological and biochemical markers for growth response
2. To assess the period of time necessary to determine the parameters which will differentiate between responders and non-responders

Inclusion criteria:

1. Ages 3 to <9 years
2. Short stature with height >2.25 Standard Deviation below the mean
3. Prepubertal (Tanner stage I) at commencement of trial
4. Peak Growth Hormone above 10ng/ml in at least one provocative test for Growth Hormone secretion
5. Signing Informed consent forms

Exclusion criteria:

1. Intra Uterine Growth Retardation
2. Growth retardation associated with malignancy, severe chronic disease, genetic syndromes and endocrine disorders
3. Diabetes
4. Treatment with any medical product which may interfere with Growth Hormone effects

Methods:

1. All participants will be treated with Growth Hormone during the first year of the study (and then in accordance with the local ethic requirement, to supply drug which is not approved for the indication used in the study, for additional 3 years) and then will be followed up for the next 3 years.
2. The impact of Growth Hormone therapy on clinical laboratory parameters that are indicative of the growth response will be assessed by collecting blood and urine samples during the 4 years study period.Samples will be test for biochemical markers of bone formation and resorption
3. The primary endpoints are measurements of height and growth velocity during the year of Growth Hormone treatment, the height at the beginning of puberty and final height. Secondary endpoints are psychological parameters, assessed by questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Ages 3 to <9 years
* Short stature with height >2.25 Standard Deviation below the mean
* Prepubertal (Tanner stage I) at commencement of trial
* Peak Growth Hormone above 10ng/ml in at least one provocative test for Growth Hormone secretion
* Signing informed consent forms

Exclusion Criteria:

* Intra Uterine Growth Retardation
* Growth retardation associated with malignancy, severe chronic disease, genetic syndromes and endocrine disorders
* Diabetes
* Treatment with any medical product which may interfere with Growth Hormone

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2006-04; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Height | every 4 months
Growth velocity | every 4 months
Height at beginning of puberty | At the biginning of puberty
Final height | When acheiving final height

SECONDARY OUTCOMES:
Psychological parameters | once a year
HbA1c and IGF-1 | at baseline. after 3 months and than every 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Phillip, Prof, MD, Principal Investigator — Schneider Children Medical Center
Locations (1):
- schneider children medical center of Israel, Petah Tikva, Israel